CLINICAL TRIAL: NCT05106829
Title: Effect of Treadmill Training Combined With Ankle Weights on Balance in Spastic Cerebral Palsied Children.
Brief Title: Treadmill With Ankle Weights on Balance in Spastic Cerebral Palsied Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Wagdy, lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003112
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy
Keywords: Treadmill; Biodex Balance System; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Physical therapy and ankle weights.
Who Masked: Participant, Outcomes Assessor
Masking Description: By random generator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy program with treadmill training without using of ankle weights. (Active Comparator): Cerebral palsied children will receive the physical therapy program from 45- 60 min./ session in addition to gait training on treadmill for 30 min./ session.
  Interventions: Other: Physical therapy program with treadmill training without using of ankle weights.
- Physical therapy program with treadmill training with using of ankle weights. (Experimental): Cerebral palsied children will receive the physical therapy program from 45- 60 min./ session in addition to gait training on treadmill with ankle weights for 30 min./ session.
  Interventions: Other: Physical therapy program with treadmill training with using of ankle weights.

INTERVENTIONS:
Other: Physical therapy program with treadmill training without using of ankle weights. — The physical therapy program include manual standing on the mat, manual standing on the mat with step forward and step backward, kneeling and half kneeling on the mat, changing position exercises from prone to standing and from supine to standing, equilibrium, protective and righting reactions using balance board and medical ball, balance training exercise from standing on the mat, strengthening exercises for weak dorsiflexors, stooping and recovery exercising from standing position, squatting to standing exercise, gait training in different directions and, stretching exercises for tight muscles (e.g: hip flexors, hamstrings and calf muscles in lower limb and for wrist flexors, pronators and elbow flexors in upper limb) + gait training on treadmill without ankle weights.
  Arms: Physical therapy program with treadmill training without using of ankle weights.
Other: Physical therapy program with treadmill training with using of ankle weights. — he physical therapy program include manual standing on the mat, manual standing on the mat with step forward and step backward, kneeling and half kneeling on the mat, changing position exercises from prone to standing and from supine to standing, equilibrium, protective and righting reactions using balance board and medical ball, balance training exercise from standing on the mat, strengthening exercises for weak dorsiflexors, stooping and recovery exercising from standing position, squatting to standing exercise, gait training in different directions and, stretching exercises for tight muscles (e.g: hip flexors, hamstrings and calf muscles in lower limb and for wrist flexors, pronators and elbow flexors in upper limb) + gait training on treadmill with ankle weights.
  Arms: Physical therapy program with treadmill training with using of ankle weights.

SUMMARY:
The purpose of the study is to investigate the effect of treadmill training combined with ankle weights on balance in spastic cerebral palsied children.

DETAILED DESCRIPTION:
Cerebral palsy defined as a non-progressive, non-hereditary lesion of the cerebral cortex resulting in postural and motion disturbances. Spastic cerebral palsied children have deficits in the selection of appropriate sensory inputs for postural control. Balance is a complex motor skill often referred to as postural control which is the ability to maintain equilibrium in a gravitational field by keeping or returning the center of body mass over the base of support. Treadmill gait training supporting the body weight which simulates walking on flat land is prescribed in rehabilitation of spastic cerebral palsy to improve their balance or to reduce their gait disturbance. Several studies support the use of ankle weights during treadmill gait training to reinforce muscle strength and, improve the symmetry of gait while, there is no research conducted on balance in spastic cerebral palsied children. Hence, there is need to study the effect of treadmill training combined with ankle weights on balance in spastic cerebral palsied children.

Fourty children with spastic hemiparetic cerebral palsied children (based on power analysis) from both sexes (6-9 years) will be recruited from different private pediatric physical therapy clinics. They will be divided randomly into control group (20 children) and study group (20 children). Control group will be participated in designed physical therapy program in addition to gait training on treadmill with full weight bearing without using of ankle weights. Study group will be participated in the same designed physical therapy program received by the control group in addition to gait training on treadmill with ankle weights on the affected side ankle.

ELIGIBILITY:
Inclusion Criteria:

1-Children ages will be ranged from 6 to 9 years old. 2-Confirmed diagnosis of hemiparetic cerebral palsy by a pediatric neurologist.

3-Spasticity grades ranged from 1 to +1 according to modified Ashworth. 4-Balance problems (frequent falling especially when increasing speed or walking on uneven surface) based on the Biodex stability system.

5-Independent standing and walking. 6-Ability to follow simple verbal commands and instructions

Exclusion Criteria:

1. Auditory or visual defects or any perceptual defects.
2. Fixed deformities on both upper or/ lower limbs.
3. Botox injection.
4. Cardiovasucular disease.
5. Surgery within the previous 24 months.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Balance | Up to 8 weeks
  Biodex Stability System will be used to measure overall stability index, anteroposterior stability index and mediolateral stability index.
Muscle strength | Up to 8 weeks
  Handheld dynamometer (Lafayette) will be used to record dorsiflexors force in pounds (Lbs)

SECONDARY OUTCOMES:
Functional balance assessment | Up to 8 weeks
  Pediatric Balance Scale will be used to assess functional balance. It contains 14 items (Sitting to standing-Standing to sitting-Transfers-Standing unsupported-Sitting unsupported-Standing with eyes closed-Standing with feet together-Standing with one foot in front-Standing on one foot-Turning 360 degrees-Turning to look behind-Retrieving object from floor-Placing alternate foot on stool-Reaching forward with outstretched arm) that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.